CLINICAL TRIAL: NCT02551601
Title: Subfoveal Choroidal Thickness in Thai Population
Status: Terminated | Type: Observational
Why Stopped: No new participants
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Yosanan Yospaiboon, Department of Ophthalmology, Faculty of Medicine, Khon Kaen University, Khon Kaen University
Other Study IDs: HE561056
Record Dates: First submitted 2015-09-15; First posted 2015-09-16 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Healthy
Keywords: subfoveal choroidal thickness; optical coherence tomography; enhanced depth imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Healthy volunteers: to measure the subfoveal choroidal thickness in healthy volunteers
  Interventions: Other: measure subfoveal choroidal thickness

INTERVENTIONS:
Other: measure subfoveal choroidal thickness — measure subfoveal choroidal thickness using optical coherence tomography

SUMMARY:
The purpose of this study was to determine the subfoveal choroidal thickness in normal Thai eyes and study the associations with gender, age, refractive error and axial length using spectral-domain optical coherence tomography with enhanced depth imaging technique.

DETAILED DESCRIPTION:
Alteration of choroidal blood supply causes changes in choroidal thickness and results in choroidal abnormalities. These are usually associated with retinal diseases and leading to severe visual dysfunction. Choroidal thickness is therefore helpful in diagnosis and treatment for many chorioretinal conditions. With the advent of spectral domain optical coherence tomography and enhanced depth imaging technique, choroidal thickness has been investigated widely in normal eyes and various chorioretinal diseases including central serous chorioretinopathy (CSC), age-related macular degeneration (AMD), highly myopia and Vogt Koyanagi-Harada disease. Similar to retinal thickness, a normal baseline choroidal thickness might be used for interpretation. This value might be affected by several variables including age, gender and ethnicity. Although there were previous studies on subfoveal choroidal thickness in normal eyes from many countries, there has been no such study in Thailand. The purpose of this study was to determine the subfoveal choroidal thickness in normal Thai eyes and study the associations with gender, age, refractive error and axial length using SD-OCT and EDI technique.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above
* Healthy subjects
* No ocular diseases
* Written informed consent form

Exclusion Criteria:

* patients with systemic diseases that may affect retinal or choroidal thickness including diabetes
* patients with history of refractive surgeries, intraocular surgeries or retinal laser treatments
* patients with history of macular, retinal, or optic nerve abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers, age 18 years or above, no ocular diseases
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
subfoveal choroidal thickness | up to 4 months
  Thickness of choroid at the foveal area

CONTACTS AND LOCATIONS:
Overall Officials: Yosanan Yospaiboon, MD, Principal Investigator — Department of Ophthalmology, Khon Kaen University
Locations (1):
- Eye outpatients department, Srinagarind Hospital, Khon Kaen University, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No